CLINICAL TRIAL: NCT02506179
Title: A Study of the Impact of Adalimumab on Patient-reported Outcomes (PROs) in Canadian Patients Suffering From Moderate-to-severe Ulcerative Colitis (UCanADA)
Brief Title: Impact of Adalimumab on Patient-reported Outcomes in Ulcerative Colitis
Acronym: UCanADA
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-325
Record Dates: First submitted 2015-06-26; First posted 2015-07-23 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
Keywords: Real-life effect; Adalimumab; Patient reported outcomes (PRO); Moderate to severe ulcerative colitis (UC); Ulcerative colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Open-label cohort: Patients will be followed for 52 weeks post initiation of adalimumab (Week 0).

SUMMARY:
To evaluate the real-life effect after 1 year of adalimumab treatment on psychological distress/depression symptoms in moderate-to-severe Ulcerative Colitis (UC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient must voluntarily sign and date a patient authorization.
* Patient must be ≥ 18 years of age.
* Patient must have confirmed diagnosis of UC.
* Patient must have:

  1. a Mayo endoscopic sub score of 2 or 3 from endoscopic investigation in the previous 3-months that is closest to the baseline visit or
  2. a Mayo rectal bleeding subscore ≥ 2 and a calprotectin value greater than 250 µg/gr.
* Patient must have been prescribed adalimumab as part of his treatment by his treating physician.
* If the patient was previously treated with vedolizumab or any anti-TNF agent (except adalimumab), an appropriate washout has taken place as per routine practice.

Exclusion Criteria:

* Patient has previously received adalimumab.
* Patient has previously used infliximab or any anti-TNF agent and have not clinically responded at any time ("primary non-responder") unless they experienced a treatment limiting reaction.
* Patient with a history of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Kock pouch, or ileostomy for UC or planned bowel surgery.
* Patient with a current diagnosis of indeterminate colitis, ulcerative proctitis only, or with a current diagnosis and/or have a history of Crohn's disease.
* Patient with other tumor necrosis factor (TNF) immune-modulated disease.
* Patient has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that in the opinion of the investigator would adversely affect his/her participating in this study.
* A female patient is pregnant or breast-feeding.
* Patient is currently participating in another prospective study including controlled clinical trials and observational studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females with moderate to severe UC patients from Canada who meet the inclusion criteria and who do not meet any of the exclusion criteria will be eligible for enrollment into the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms at Week 52 | From Week 0 to Week 52 or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  It is measured by the Patient Health Questionnaire - 9 Items (PHQ-9).

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms at Week 8 | From Week 0 to Week 8, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  It is measured by the Patient Health Questionnaire - 9 Items (PHQ-9).
Change from baseline in the proportion of patients with PHQ-9 >= 10 | From Week 0 to Week 52 or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  The change from baseline in the proportion of patients with PHQ-9 >= 10 is assessed at week 8 and 52.
Change from baseline in Disability | From Week 0 to Week 52 or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  It is measured by the Inflammatory Bowel Disease (IBD) Disability Index at weeks 8 and 52.
Change from baseline in Overall quality of life | From Week 0 to Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  It is measured by the EuroQol 5-Dimensions, 5 Levels (EQ-5D-5L) and EQ5D VAS at weeks 8 and 52.
Change from baseline in Ulcerative Colitis (UC)-specific quality of life | From Week 0 to Week 52 or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  It is measured by the Short Quality of Life in Inflammatory Bowel Disease Questionnaire (SIBDQ) at weeks 8 and 52.
Change from baseline in Fatigue | From Week 0 to Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  It is measured by the Functional Assessment Chronic Illness Therapy-Fatigue (FACIT-F) at weeks 8 and 52.
Change from baseline in Sleep impairment, | From Week 0 to Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  It is measured by the Medical Outcomes Study Sleep scale (MOS Sleep) at weeks 8 and 52.
Change from baseline in Work productivity | From Week 0 to Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  The change from baseline in work productivity is assessed at week 8 and 52.
Assessing Simple Clinical Colitis Activity Index (SCCAI) | Up to Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  SCCAI is used to access response and remission rates.
Change from baseline in Fecal Calprotectin levels | From Week 0 to Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  The change from baseline in Fecal Calprotectin levels will be assessed.
Mayo endoscopic sub-score | Up to Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  Mayo endoscopic sub-score will be assessed.
Proportion of patients with Complications including hospitalization and surgery | At Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  The proportion of patients with complications including hospitalization and surgery will be assessed.
Proportion of patients on steroids | At Week 52, or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  The proportion of patients on steroids will be assessed.
Change from baseline in Physician's Global Assessment (PGA) | From Week 0 to Week 52 or at the time of stopping adalimumab, or at the time of Premature Discontinuation
  The change from baseline in Physician's Global Assessment (PGA) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (23):
- Canada (23):
  - University of Calgary /ID# 144032, Calgary, Alberta
  - Zeidler Ledcor Centre /ID# 145973, Edmonton, Alberta
  - Columbia Gastro Mgmnt Ltd /ID# 136820, New Westminster, British Columbia
  - GIRI Gastrointestinal Research Institute /ID# 141107, Vancouver, British Columbia
  - Discovery Clinical Services /ID# 144102, Victoria, British Columbia
  - Percuro Clinical Research, Ltd /ID# 136533, Victoria, British Columbia
  - Dr. Everett Chalmers Reg Hosp. /ID# 136534, Fredericton, New Brunswick
  - Dr Chadwick Ian Williams Professional Corporation /ID# 144802, Saint John, New Brunswick
  - Bellini Medicine Professional /ID# 144241, Brampton, Ontario
  - Oshawa Clinic /ID# 144364, Oshawa, Ontario
  - The Ottawa Hospital /ID# 139392, Ottawa, Ontario
  - Kensington Screening Clinic /ID# 141106, Toronto, Ontario
  - Mount Sinai Hosp.-Toronto /ID# 141108, Toronto, Ontario
  - Dr O Tarabain Medicine Prof Corp /ID# 144034, Windsor, Ontario
  - Dr. Rahman Bacchus Med. Corp. /ID# 141780, Windsor, Ontario
  - Hopital Hotel-Dieu de Levis /ID# 137099, Lévis, Quebec
  - Hospital Maisonneuve-Rosemont /ID# 137336, Montreal, Quebec
  - CHUM - Hopital Saint-Luc /ID# 139393, Montreal, Quebec
  - McGill Univ HC /ID# 136821, Montreal, Quebec
  - Clinique MEDI-CLE /ID# 153690, Montreal, Quebec
  - CHU de Quebec-Universite Laval /ID# 147557, Québec, Quebec
  - CHUS - Hopital Fleurimont /ID# 137840, Sherbrooke, Quebec
  - Royal Univ. Hosp, Saskatoon,CA /ID# 137838, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P15-325.pdf